CLINICAL TRIAL: NCT03488043
Title: Predictive Score of PneumOThorax Secondary to CT-guided Transthoracic Lung Biopsy Made From a Large Retrospective Cohort and Validated on a Prospective Cohort
Acronym: SPOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/372
Record Dates: First submitted 2018-03-26; First posted 2018-04-04 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-03

CONDITIONS: Pneumothorax
Keywords: Lung lesions; Pneumothorax; CT-guided transthoracic biopsy; Risk score
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: All patients having a CT-guided transthoracic biopsy from September 2012 and September 2017.
  Interventions: Procedure: Needle lung biopsy
- Prospective cohort: All patients having a CT-guided transthoracic biopsy from April 2018.
  Interventions: Procedure: Needle lung biopsy

INTERVENTIONS:
Procedure: Needle lung biopsy — Needle lung biopsy

SUMMARY:
Transthoracic lung biopsy (TLB) provides a histological diagnosis of nodule or lung mass. Pneumothorax is the main complication of TLB with an average of 20%. Many risk factors, whether clinical, computed tomography or related to TLB, are described in the literature. The British Thoracic Society recommends monitoring for 2 hours after the procedure with a possible discharge if the chest X-ray is normal. There is no French or European recommendation for monitoring the occurrence of pneumothorax after TLB. In the university center of Besançon, France, a minimum supervision of 4 hours is recommended and approximately one in two patients is hospitalized until the following day to reach this minimum time of 4 hours. The objective of the SPOT study is to perform a predictive score of pneumothorax from a retrospective cohort of patients for whom a transthoracic lung biopsy was performed and to validate this score on a prospective cohort. The expected goal is to select patients who can benefit from outpatient care by shortening the post-procedure surveillance period and to monitor more long-term only high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients having needle lung biopsy CT-guided for diagnostic purposes.

Exclusion Criteria:

* Nodule or mass in contact with the pleura for which the aerated pulmonary parenchyma is not crossed by the puncture needle.
* Several pulmonary sites biopsied.
* Existence of a pneumothorax before procedure
* Per-procedural appearance of alveolar or interstitial pneumonitis at the level of the biopsy area.
* Cavitary aspect of nodule or mass
* Absence of chest X-ray control
* Poorness quality of chest X-ray control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See eligibilty criteria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Pneumothorax occurrence | between 4 and 24 hours after procedure
  Pneumothorax is defined by the observation on the chest x-ray of a pleural detachment regardless of its importance.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lamfichekh Y, Lafay V, Hamam J, Guillien A, Puyraveau M, Behr J, Manzoni P, Calame P, Dalphin JC, Eberst G, Grillet F, Westeel V. Score to Predict the Occurrence of Pneumothorax After Computed Tomography-guided Percutaneous Transthoracic Lung Biopsy. J Thorac Imaging. 2023 Sep 1;38(5):315-324. doi: 10.1097/RTI.0000000000000729. Epub 2023 Jul 17. PMID 37603106